CLINICAL TRIAL: NCT05265455
Title: Randomized Clinical Trial, Controlled Against Placebo, Performed to Evaluate the Effect of a Phytosterol-based Product (2.5 g/Day), After 3 Weeks of Intake, on the Lipid Profile, Also in Relation to the Quality of the Diet, in Subjects With Moderate Hypercholesterolemia and Low / Moderate Global Cardiovascular Risk
Brief Title: Diet and Plant Sterols in the Control of Cholesterolemia (DESCO)
Acronym: DESCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Professor, University of Bologna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DESCO_2021
Record Dates: First submitted 2021-11-24; First posted 2022-03-03 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Phytosterols

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant sterol supplementation (Experimental): 2.5 g of phytosterols in pre-dosed sticks (oral supplementation)
  Interventions: Dietary Supplement: Plant sterols 2.5 g/day
- Placebo (Placebo Comparator): Placebo in pre-dosed sticks (the same matrix without plant sterols) (oral supplementation)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plant sterols 2.5 g/day — Daily consumption of one stick (2.5 g of plant sterols) during lunch or dinner for 3 weeks
  Arms: Plant sterol supplementation
Dietary Supplement: Placebo — Daily consumption of one stick (the same matrix without plant sterols) during lunch or dinner for 3 weeks
  Arms: Placebo

SUMMARY:
DESCO is a randomized clinical trial, controlled against placebo, performed to evaluate the effect of a phytosterol-based product (2.5 g/day), after 3 weeks of intake, on the lipid profile, also in relation to the quality of the diet, in subjects with moderate hypercholesterolemia and low / moderate global cardiovascular risk.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, monocentric cross over clinical study conducted in Italy.

The objective of this study is to evaluate the fasting lipid profile of adults with moderate hypercholesterolemia and a low/very low cardiovascular risk, after 3 weeks of supplementation with 2.5 g/day of plant sterols, vs placebo, and to assess the relationship between the effects of the supplementation and the diet.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol plasma levels between 200 and 240 mg/dL and/or LDL cholesterol levels between 130 and 160 mg/dL
* Triglyceride plasma levels <200 mg / dL
* Cardiovascular risk at 10 years (according to the SCORE algorithm) <5%.
* Signature of the informed consent form

Exclusion Criteria:

* Subjects in secondary prevention for cardiovascular diseases or with a global cardiovascular risk (according to the SCORE algorithm) > 5% at 10 years
* Triglyceride plasma levels >200 mg / dL
* Decompensated diabetes
* Alcoholism
* Food allergy
* Recent intake of functional foods or supplements for cholesterol control
* Intake of lipid-lowering drugs or drugs affecting lipid metabolism in the last 2 months
* Alterations in thyroid, hepatic or renal function (transaminases greater than 3 times the maximum values; glomerular filtration rate <30ml / min), muscle diseases, even if subclinical
* Obesity (BMI> 30)
* Any medical or surgical condition that could make the patient's adherence to the study protocol complex or inconstant.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Fasting lipid profile | 3 weeks
  Evaluation of the effects of the intake of phytosterols on fasting lipid profile, including the following parameters: total and LDL cholesterol, triglycerides, HDL cholesterol, plasma levels of apolipoproteinB-100.

SECONDARY OUTCOMES:
Mediterranean index of the diet assessed by validated FFQ | 3 weeks
  Assessment of the relationship between the effects of the supplementation with phytosterols and the Mediterranean index of the diet assessed by using a validated food frequency questionnaire (Gnagnarella et al. Nutr Metab Cardiovasc Dis. 2018;28:1140-1147).
Weight | 3 weeks
  Evaluation of the effects of the intake of phytosterols on weight in kilograms
BMI | 3 weeks
  Evaluation of the effects of the intake of phytosterols on BMI (weight kilograms and height meters will be combined to report BMI in kg/m^2 )
Abdominal circumference | 3 weeks
  Evaluation of the effects of the intake of phytosterols on abdominal circumference
Blood pressure | 3 weeks
  Evaluation of the effects of the intake of phytosterols on blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cicero AFG, Fogacci F, Giovannini M, Rizzoli E, Grandi E, D'Addato S, Borghi C. The Effect of Dietary Supplementation with Plant Sterols on Total and LDL-Cholesterol in Plasma Is Affected by Adherence to Mediterranean Diet: Insights from the DESCO Randomized Clinical Study. Nutrients. 2023 Oct 27;15(21):4555. doi: 10.3390/nu15214555. PMID 37960208